CLINICAL TRIAL: NCT02667990
Title: Maximal Plantar Pressure and Comfort Evaluation During Normal Every Day Use of an "Orthopedic" Stiletto, a Normal Stiletto and a Control Trainer Shoe
Brief Title: Maximal Plantar Pressure and Comfort Evaluation of Orthopedic Stilettos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Jeannette Penny, orthopedic surgeon, PhD., Copenhagen University Hospital, Hvidovre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 47798
Record Dates: First submitted 2015-08-28; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Metatarsalgia
Keywords: metatarsalgia; pedobar; foot; stiletto; insoles
MeSH Terms: conditions — Metatarsalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- orthopaedic stilettoe (Experimental): orthopaedic stilettoe will be compared to standard stilettoe and comfy trainer
  Interventions: Other: orthopaedic stilettoe; Other: standard stiletto; Other: comfy trainer

INTERVENTIONS:
Other: orthopaedic stilettoe — stilettos with orthopaedic in-sole buildt into the shoe
Other: standard stiletto — standard stiletto without insole
Other: comfy trainer — comfy trainer

SUMMARY:
22 women Testing "orthopedic" stilettos compared to standard stilettos and a comfy trainer.

Testing involves pedobar pressures and a validated comfort questionnaire.

DETAILED DESCRIPTION:
22 women Testing "orthopedic" stilettos compared to standard stilettos and a comfy trainer testing involved pedobar pressures and a validated comfort questionnaire.

x rays with arthrosis 1. metatarsophalangeal joint (MTPJ), hallux valgus and Intermetatarsal (IM) angles will be recorded.

Clinically, weight, height, foot length, heel valgus, 1. MTPJ range of motion, pain, callus, hammertoes will be recorded.

Sole pressure in heel, arch and forefoot grids measured by in-sole pressure pedar-x (Novel) and possible Emed system (Novel).

3 working days in each type of shoe with Steps measured by pedometer Comfort assed as VAS according to: Mundermann,A., Nigg,B.M., Stefanyshyn,D.J., and Humble,R.N.: Development of a reliable method to asses footwear comfort during running. Gait Posture, 16:38-45, 2002.

Primary outcome is the foot sole pressures. Both VAS comfort and foot pressures will be regressed to see if age, BMI, shoe size, steps, shoe type, callus, index minus, hallux valgus etc has an effect.

16 needed for the pressure and 21 for the comfort score. 22 will be included to make sure the investigators have enough power.

ELIGIBILITY:
Inclusion Criteria:

* Foot healthy females used to wearing stilettos.

Exclusion Criteria:

* Shoe sized outside European 37-42.
* Sought doctor for foot or balance related issues

Ages: 18 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
plantar foot pressure | 1 hrs
  Mean and peak pressure and pressure/time in the heel, arch and fore foot ( fore foot subdivided into 1. metatarsal head, 2+3 rd head, 4+5th head and the big toe). Pressure measured as Newton/sq. cm.

SECONDARY OUTCOMES:
comfort rating footwear | 1 month
  VAS scale indication comfort around the shoe. The scale is continuous from 0 to 15, with 15 being the most comfortable condition imaginable. It measures: Overall comfort, Heel cushioning, Forefoot cushioning, Arch height, Heel cup fit, Heel cup width, Shoe forefoot width, Shoe length. The investigators will register all but the overall comfort and the cushioning measures are assumed the most interesting measures in this study. (Mundermann,A., Nigg,B.M., Stefanyshyn,D.J., and Humble,R.N.: Development of a reliable method to assess footwear comfort during running. Gait Posture, 16:38-45, 2002.)

OTHER OUTCOMES:
X ray angles of the foot | 1 hrs
  Hallux valgus, Intermetatarsal and O'Meary angles, index minus (Rui Baracco 2011) and signs of arthrosis (Cockhlin 2003 grade 0-4)

CONTACTS AND LOCATIONS:
Overall Officials: jeannette penny, PhD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Hvidovre Hospital, Hvidovre, Denmark